CLINICAL TRIAL: NCT07243405
Title: The Evaluation of Neuro Stimulation for Treatment of Sleep Disordered Breathing
Brief Title: Neurostimulation for Sleep Disordered Breathing (SDB)
Acronym: ECLIPSE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lunair Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10138
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disordered Breathing (SDB); Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, single arm, feasibility clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpha Lunair System implanted subjects (Experimental)
  Interventions: Device: Neuro stimulator implant

INTERVENTIONS:
Device: Neuro stimulator implant — Neuro stimulator for treating sleep disordered breathing

SUMMARY:
This is a study to determine if the Lunair Alpha System is safe and effective for treating moderate to severe sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Subject does not tolerate, not compliant to, or have access to alternative Sleep Disordered Breathing treatments
* Subject has moderate to severe sleep disordered breathing as diagnosed by PSG

Exclusion Criteria:

* Subject is taking opioids, narcotics, sleep or psychotic medications or supplements that may alter consciousness, the pattern of respiration, sleep architecture, or with known effect on sleep-wake function or alertness.
* Any reason for which, in the judgement of the investigator, the subject is considered to be a poor study candidate
* Subject has previous upper respiratory tract (URT) surgery or procedure (e.g., uvula, soft palate or tonsils) within 60 days prior to Screening PSG.
* Subject has a need for chronic supplemental oxygen therapy for any reason
* Subject has other sleep disorders or sleep hygiene behaviors that confound functional assessments of sleepiness
* Subject has severe chronic kidney disease
* Subject exhibits ongoing misuse of alcohol, tobacco, caffeine, or recreational drugs that would impact either the results of or the participation in a sleep study
* Subject conducts work or regular activities requiring vigilance
* Subject is unwilling or unable to refrain from consumption of alcoholic beverages for 24 hours prior to the start of each PSG study
* Subject is unwilling or unable to refrain from sleep disordered breathing treatments or devices
* Subject has an active systemic infection at the time of implant
* Subject has clinical evidence of immunodeficiency
* Any condition likely to require future MRI or diathermy
* Subject is pregnant
* Subject has severe nasal obstruction that could restrict airflow
* Subject has any trauma to the upper airway
* Subject has previous surgical resection, prior or current radiation therapy for cancer or congenital malformations in the larynx, tongue, or throat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - assessment of procedure or device related adverse events | enrollment to 12 months post-implant
  Incidence of adverse events (AEs) related to the Lunair system or procedure

SECONDARY OUTCOMES:
Improvement in sleep disordered breathing per sleep study | six month, 12 month and 24 month post implant
  Improvement in sleep disordered breathing at 6,12 and 24 months post implant during an attended sleep study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Paitilla, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No